CLINICAL TRIAL: NCT00460785
Title: Phase 1 Single Center Trial to Demonstrate the Bioequivalence of a New Combination Analgesic Formulation as Compared to an Equimolar Marketed Formulation
Brief Title: Bioequivalence Trial of a New Opioid Combination Compared to Reference
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 544506
Record Dates: First submitted 2007-03-28; First posted 2007-04-16 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-03

CONDITIONS: Healthy
MeSH Terms: interventions — Analgesics, Opioid

INTERVENTIONS:
Drug: Opioid

SUMMARY:
The purpose of this study is to demonstrate bioequivalence of a new formulation to a reference

ELIGIBILITY:
Inclusion Criteria:

* Standard Phase I
* Cyp 2D6 extensive metabolizers

Exclusion Criteria:

* Standard Phase I
* Contraindications of current reference tablet SmPC

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2007-02; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence acceptance range of 90CI of T/R ratios of AUC and Cmax.

SECONDARY OUTCOMES:
Descriptive, e. g. safety/tolerability of Test comparable to Reference

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Timmer, Dr., Principal Investigator — CRS Mannheim